CLINICAL TRIAL: NCT06746259
Title: CLP-0019- FebriDx® Method Comparison Study Protocol
Brief Title: FebriDx® Method Comparison Study Protocol
Status: Completed | Type: Observational
Sponsor: Lumos Diagnostics (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CLP-0019
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: Point of care diagnostics; CRP (C- Reactive Protein); MxA (Myxovirus resistance protein A)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Untrained Operator: Untrained Operators have no training or hands-on experience in conducting laboratory testing (moderate or high complexity). Should not have previous training or experience with FebriDx but may have limited experience with other waived or home use tests.
  Untrained operators will test patients with ARI with the FebriDx test after reviewing and familiarizing themselves with the study articles and the manufacturer's instructions (QRI and IFU).
  Interventions: Diagnostic Test: Rapid point of care test to detect host immune response in ARI
- Trained Operator: Trained operators are qualified to perform moderate complexity testing and have previous training and/or experience with the FebriDx test.
  Trained operators will test patients with ARI with the FebriDx test after completing a training seminar which includes review of the test procedure as described in the IFU/QRI, a competency test, interpretation of mock test results, as well as at least one (1) practice test
  Interventions: Diagnostic Test: Rapid point of care test to detect host immune response in ARI

INTERVENTIONS:
Diagnostic Test: Rapid point of care test to detect host immune response in ARI — FebriDx is a rapid lateral flow immunoassay for the visual, qualitative, in vitro detection of elevated levels of host response proteins, Myxovirus resistance protein A (MxA) and C-reactive protein (CRP), directly from fingerstick blood to aid in the differentiation of bacterial from non-bacterial acute respiratory infections.
  Other Names: Fingerstick test

SUMMARY:
The goal of this observational study is to learn about the performance and ease of use of FebriDx when operated by persons without laboratory experience or training in patients with acute respiratory symptoms. The main question it aims to answer is:

• Is FebriDx accurate at differentiating bacterial from non-bacterial respiratory infections when used by untrained operators? Trained and untrained participants will run the FebriDx test on patients with respiratory symptoms to evaluate comparability.

DETAILED DESCRIPTION:
A prospective, multi-center, blinded observational study to demonstrate that the FebriDx test meets the CLIA statutory criteria for waiver by providing sufficient assurance that the addition of a new operator population (untrained) and environment of use (waived) will not adversely impact the performance or safety of the test.

The study aims to:

* Demonstrate that FebriDx® Test is accurate and the operator can perform the test with a negligible risk of erroneous result.
* As a secondary objective, ease-of-use objective data and subjective feedback relating to the device and its operator interface will be collected at the end of the study and assessed for comparability.

ELIGIBILITY:
Inclusion Criteria:

* Subject exhibits or reports a new onset measured temperature (oral or tympanic) of greater than or equal to 100.5°F/38°C within 3 days (72 hours) of enrollment or at the visit
* Subject has clinical suspicion for Acute Respiratory Infection and presents with at least one (1) of the following new onset symptoms beginning ≤ 7 days of enrollment: runny nose, nasal congestion, sore throat, cough, hoarse voice or shortness of breath

Exclusion Criteria:

* Subject is unable or unwilling to provide signed, Informed Consent
* Subject is less than 12 years old or over 64 years old
* Subject has a fever that started more than 3 days (> 72 hours) prior to enrollment
* Subject has symptoms of Acute Respiratory Infection that started > 7 days of enrollment
* Subject is receiving interferon therapy (e.g. MS, HIV, HBV, HCV) in the last 30 days
* Subject is in an immunocompromised state (e.g. HIV) or taking immunosuppressive or chemotherapeutic medications in the last 30 days (e.g. oral steroids, Methotrexate, Cyclosporine, Antimetabolite chemotherapy, interferon therapy)
* Subject has taken antibiotics or antiviral therapy in the last 14 days
* Subject received a live viral immunization in the last 14 days
* Subject has significant trauma or burns (> 5% total body surface area or full thickness (3rd°)) in the last 30 days
* Subject has had major surgery (requiring intravenous anesthesia and/or respiratory assistance) in the last 30 days
* Subject has a history of a myocardial infarction or stroke in the last 30 days

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Symptomatic patients presenting to outpatient settings (e.g., physician offices, clinics, urgent care centers) with recent fever (reported within the last 72h) and recent symptoms of acute respiratory infection (symptoms reported to have started ≤ 7 days prior to study visit).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Performance | Day 1
  Positive Percent Agreement (PPA), Negative Percent Agreement (NPA) and 95% confidence intervals will be calculated for each untrained operator and compared to performance in trained operators (truth).

SECONDARY OUTCOMES:
Usability | Day 1
  Ease-of-use objective data and subjective feedback relating to the device and its Operator interface will be collected at the end of the study

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Ascada Health, Fullerton, California
  - Exer Urgent Care, Pasadena, California
  - L&C, Miami, Florida
  - Trujillo Medical Center, Miramar, Florida
  - Hillcrest Medical Research, LLC, Orange City, Florida
  - Hometown Urgent Care and Research, Beavercreek, Ohio
  - HMG Clinical Research/Herrera Medical Group, Bedford, Texas
  - Ascada Health, Katy, Texas